CLINICAL TRIAL: NCT03424980
Title: A Real-world Non-interventional Observational Study to Evaluate Effectiveness and Safety of Tyrosine Kinase Inhibitors (TKIs) in the Patients With Non-small Cell Lung Cancer Complicated With Brain Metastases
Brief Title: A Study to Evaluate Effectiveness and Safety of Tyrosine Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhang Helong, Professor, Tang-Du Hospital
Other Study IDs: W-TONG03
Record Dates: First submitted 2018-01-18; First posted 2018-02-07 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Non-small cell lung cancer, Chinese, brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tyrosine kinase inhibitors: Diagnosed patients with advanced non-small cell lung cancer (NSCLC) with brain metastases who were administered with tyrosine kinase inhibitors only or combination therapies of tyrosine kinase inhibitors
  Interventions: Combination Product: Tyrosine kinase inhibitors

INTERVENTIONS:
Combination Product: Tyrosine kinase inhibitors — Tyrosine kinase inhibitors only or combinations therapies of tyrosine kinase inhibitors

SUMMARY:
This is a real-world non-interventional observational study. The study was designed to evaluate the effectiveness and safety of clinical treatments in the patients with advanced non-small cell lung cancer (NSCLC) complicated with brain metastases in clinical practice.

DETAILED DESCRIPTION:
This is a real-world non-interventional observational study that focuses to evaluate the effectiveness and safety of tyrosine kinase inhibitors (TKIs) in the patients of advanced non-small cell lung cancer (NSCLC) with brain metastases diagnosed by medical imaging methods. The patients with core medical health records who were enrolled in the clinics from 2014 to 2017 and were administered with TKIs only or combination therapies of TKIs will be included in the study. All the treatments followed real-world clinical practices and experiences of clinical physicians.

The effectiveness will be measured by the treatment effects on brain metastases (objective remission rate) and overall survival/progress-free survival. The safety will be evaluated by adverse events, serious adverse events, laboratory tests, electrocardiogram, vital sign, and physical examination. The mutation status of epidermal growth factor receptor (EGFR) and the type of anaplastic lymphoma kinase (ALK) will be assessed. All the study procedures will be in compliance with International Clinical Harmonization - Good Clinical Practice (ICH-GCP), standard operation procedures (SOPs), and regulatory policies/regulations.

ELIGIBILITY:
Inclusion Criteria:

* The patients were treated with lung cancer and were enrolled from Jan 2013 to Jun 2017
* The patients with advanced (Clinical stage: Phase IV) non-small cell lung cancer who have complete core health medical records (HMRs);
* The patients who are observed with brain metastases diagnosed by imaging methods;
* The patients who have complete clinical data for diagnosis time of brain metastases, and overall survival/effectiveness;
* The patients who are administered with tyrosine kinase inhibitors only or combination therapies of tyrosine kinase inhibitors;

Exclusion Criteria:

No exclusion criteria are included in the study given that the study is designed as non-interventional and all the treatments followed real-world clinical practice and experiences of clinical physicians.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The target study population is defined as the patients who were diagnosed with advanced non-small cell lung cancer (NSCLC) with brain metastases and were treated with tyrosine kinase inhibitors only or combination therapies of tyrosine kinase inhibitors following real-world clinical practice and experiences of clinical physicians
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who are not observed with the event of objective remission | 2013 - 2017
  Percentage of patients who are not observed with the event of objective remission

SECONDARY OUTCOMES:
Percentage of patients who are not observed with the event of disease progression | 2013 - 2017
  Percentage of patients who are not observed with the event of disease progression

OTHER OUTCOMES:
Percentage of patients who are not observed with the event of overall survival | 2013 - 2017
  Percentage of patients who are not observed with the event of overall survival
Percentage of patients with adverse events and serious adverse events | 2013 - 2017
  Percentages of patients with adverse events and serious adverse events (Percentages of the numbers of reported adverse events/total population * 100%)
Severity of adverse events | 2013 - 2017
  Severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, Principal Investigator — Xi'an Tangdu Hospital
Locations (5):
- China (5):
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No